CLINICAL TRIAL: NCT04779983
Title: Evaluation of Professional Practices in the Prescription of Biological Treatments for RA Taking Into Account IL6 as a Biomarker
Brief Title: IL-6 as a Biomarker for Personalized Treatment of PR
Acronym: REMISIX
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0100
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
Keywords: IL-6; Biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several studies have shown the relevance of the IL6 level before treatment or after 6 months, as a predictive biomarker for the persistence of remission. The IL6 assay is now routinely available using the instruments available at the Montpellier University Hospital and with reagents provided by the ROCHE Laboratory. Moreover medical practices should incorporate this parameter. However, relevant threshold shlould be defined before being able to integrate biomarkers such as IL6 for monitoring bDMARDs in an algorithm.

The medical staff of Clinical Immunology Unit has decided to include the dosage of IL-6 during a routine biological assessment during patient visit to follow the new EULAR recommendations . This measument will be perfom in addition to the CRP and biochemical parameters on subjects with active RA or in remission upon the introduction of biological treatments or JAKi or during remission after at least 6 months of treatment. From March to July 2021, 200 patients will beenrolled and will benefit of this assessement. The investigators will retrospectively define clinical correlations with serum IL6 levels in order to define a threshold. In the second stage, a decisional algorithm based on the results of this project will be create. This will allow an improvement of the medical practices thanks to the integrationof of serum IL6 dosage as a standard during patients visits. The IL-6 assay will be performed on the e801 module of the Cobas lines (Roche Diagnostics) currently in place in the Biochemistry and Hormonology laboratory. The Elecsys® IL-6 - Roche Diagnostics test, high sensitivity, is an electrochemiluminescence immunoassay.

ELIGIBILITY:
Inclusion criteria:

* 18 to 65 years old
* patients with rheumatoid arthritis according to 2010 ACR/EULAR criteria who have one of the following conditions:

  * Subjects with active RA (DAS28> 3.6) who have failed methotrexate treatement and with a standard medical care for which an indication for biotherapy is retained or
  * Subjects with remission of RA (DAS28<2.6) for which a biotherapy delay (anti-TNF or anti-IL6R or JAKi) is proposed.

Exclusion criteria:

- Age under 18 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with active RA (DAS28> 3.6) who have failed methotrexate treatement and with a standard medical care for which an indication for biotherapy is retained.
  Subjects with remission of RA (DAS28<2.6) for which a biotherapy delay (anti-TNF or anti-IL6R or JAKi) is proposed.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
serum IL6 levels. | 1 day
  serum IL6 levels. From first COVID-19 symtpoms, or first positive SARS-COV2 PCR result, to recovery.

SECONDARY OUTCOMES:
The clinical correlations das 28 with the serum IL6 level | 1 day
  The clinical correlations das 28 with the serum IL6 level

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jorgensen, PU PH, Study Director — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC